CLINICAL TRIAL: NCT06123481
Title: Autologous Bone Marrow Aspirate Concentrate for the Treatment of Osteonecrosis of the Femoral Head
Brief Title: Autologous Bone Marrow Aspirate Treatment for Early-Stage Osteonecrosis
Acronym: BATON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00289774; U01AR080993-01A1 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-11-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Osteonecrosis of the Femoral Head; Avascular Necrosis of the Femoral Head
Keywords: osteonecrosis; aseptic necrosis; avascular necrosis (AVN); bone marrow aspirate; bone marrow aspirate concentrate; bone marrow cells; bone marrow; cell-based treatment; core decompression; femoral head; necrosis; bone diseases; musculoskeletal diseases; pathologic processes; hip; ONFH; AVN
MeSH Terms: conditions — Legg-Calve-Perthes Disease; Femur Head Necrosis; Osteonecrosis; Necrosis; Bone Diseases; Musculoskeletal Diseases; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: A 1:1 randomized, parallel design with two treatment arms: 1) core decompression (percutaneous drilling) alone, or 2) core decompression augmented with autogenous bone marrow aspirate. Cluster randomization will be performed at each participating institution.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded as to group assignment. Both groups will undergo a core decompression. One group will undergo a bone marrow aspiration and the other group will undergo a sham procedure. This sham procedure consists of a small incision and placing a needle up to the iliac bone but with no bone penetration or aspiration.
  The study radiologists will be blinded as to patient treatment assignment; images will be assigned the patient study number and date only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core decompression (CD) (Active Comparator): Core decompression of the femoral head with sham bone marrow aspiration
  Interventions: Procedure: Core Decompression
- Bone Marrow Aspirate Concentrate (BMAC) (Experimental): Autologous bone marrow aspiration is concentrated and injected into the necrotic bone of the femoral head through the core decompression opening.
  Interventions: Procedure: Core Decompression; Procedure: Core Decompression Procedure with Autologous Bone Marrow Aspirate Concentrate

INTERVENTIONS:
Procedure: Core Decompression — Standard core decompression procedure is performed by drilling into the necrotic bone of the femoral head. A sham bone marrow aspiration involves advancing a needle to the iliac crest (no bone penetration, no bone marrow aspiration) through a small skin incision.
Procedure: Core Decompression Procedure with Autologous Bone Marrow Aspirate Concentrate — This involves bone marrow aspiration, concentrating the bone marrow aspirate, and injecting 6 milliliters of bone marrow aspirate concentrate into the necrotic femoral head through an opening created by the core decompression.
  Arms: Bone Marrow Aspirate Concentrate (BMAC)

SUMMARY:
Osteonecrosis of the femoral head (ONFH) is a debilitating musculoskeletal disease that is characterized by localized death of bone cells and associated cellular elements within the subchondral bone. If it progresses, it results in the collapse of the femoral head (ball part of the hip) giving rise to secondary arthritis. This condition is associated with marked pain and loss of function, often necessitating a joint replacement. Due to the relatively young age of onset of ONFH (often in 20s and 30s), there is great interest in utilizing joint-preserving procedures prior to the need for joint replacement. Joint-preserving procedures include core decompression (CD) with and without bone grafts or cells, vascularized and non-vascularized bone grafting, as well as osteotomies. Inconsistent results for each of these procedures have been reported and there are no Clinical Practice Guidelines or medical community consensus opinions regarding the treatment of early-stage ONFH. The hypothesis to be tested is "Participants who have early-stage ONFH undergoing CD augmented with autogenous bone marrow aspirate concentrate will have better clinical and radiological outcomes than CD alone." This multi-center randomized controlled trial for early-stage ONFH is prospective and controlled for participant stage (only early-stage pre-collapse individuals) and surgical technique. Participants will be evaluated as per routine surgical follow-up, and at 6 months (telemedicine), 1- and 2- years using radiographs, MRIs, and questionnaires. This project will also explore the scientific basis for success vs. failure in individuals who have osteonecrosis, and have different demographics and bone marrow aspirate cell profiles.

DETAILED DESCRIPTION:
Rationale. It is estimated that there are 10,000 to 20,000 new cases of osteonecrosis of the femoral head diagnosed each year in the United States. Several approaches to treatment have been undertaken including nonsurgical (e.g., pharmaceuticals, hyperbaric oxygen) and surgical (e.g., core decompression, bone grafting (both non-vascularized and vascularized), osteotomies, total joint replacement). Total joint replacement is performed to treat end-stage disease (when the joint goes "out-of-round", and cartilage damage has occurred). There has been increasing interest in using cell-based treatment with core decompression (CD) to treat early-stage osteonecrosis. Bone marrow aspirate concentrate (BMAC) injected into the CD is being evaluated in this study as it contains progenitor cells and other elements that have been shown to facilitate the development of bone and blood vessels. There is a need for rigorous, randomized controlled studies to determine the effectiveness of this cell-based treatment for osteonecrosis of the femoral head (ONFH).

Objectives. The goal of this study is to compare the clinical and radiological results of core decompression with autologous bone marrow aspirate concentrate to core decompression alone (CD). The results will be based on: 1) evidence of radiological progression of ONFH, 2) time to radiological progression of ONFH to Association Research Circulation Osseous (ARCO) Stage III or IV, Association Research Circulation Osseous (ARC)), the international society for the study of osteonecrosis and other disorders of bone circulation] or 3) pain requiring surgical intervention. Success will be based on survivorship of the femoral head over the course of the study. Failure of the procedure is based upon evidence of radiographic progression to ARCO Stage III or pain requiring a surgical intervention.

Overall Design. This is a prospective, multi-center, interventional clinical trial being conducted to evaluate two treatments for early stage ONFH. Participants will be 1:1 randomized to one of two arms: 1) BMAC: Core decompression augmented with autogenous bone marrow aspirate concentrate; 2) CD: Core decompression alone. The core decompression and bone marrow aspiration and concentration will be performed according to a standardized protocol. The CD group will also undergo a sham procedure consisting of a small incision and placing the needle up to the iliac bone without marrow aspiration. In the BMAC group, a sample of the bone marrow aspirate concentrate will be submitted for laboratory assessments to identify the constituent cells and major biological pathways involved. Clinical Research Forms (pre-operatively; 6-, 12-, and 24-months post-operatively), radiographs, and MRIs (pre-operatively; 12- and 24-months post-operatively) will be performed.

ELIGIBILITY:
Inclusion Criteria

* Participants who have non-traumatic osteonecrosis of the femoral head
* Only participants who have Stage 1 or 2 osteonecrosis as assessed by the 2019 ARCO Staging System
* No evidence of subchondral fracture
* All osteonecrotic lesion sizes
* All major risk factors (e.g. corticosteroids, alcohol, organ recipient) except for those listed in the exclusion criteria
* Participants diagnosed who have femoral head osteonecrosis for which no risk factor has yet to be identified
* Participants will include all ethnicities and races
* Be able and willing to participate in study and return for postoperative visits

Exclusion Criteria

* Participants who have:

  * Sickle Cell disease
  * Major trauma
  * Post-irradiation ON
  * Gaucher Disease
  * Juvenile form: Legg-Calve-Perthes Disease
  * Juvenile form: Spontaneous ON of the hip
  * Pregnant or breastfeeding
  * Vulnerable population; i.e., prisoners and institutionalized individuals
* Participant is unable to undergo an MRI
* Participants who have evidence of a subchondral fracture
* Prior history of hip surgery, more extensive than hip arthroscopy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Radiological progression of osteonecrosis of the femoral head (ONFH) to ARCO Stage III or IV | Up to 24 months
  The 2019 ARCO Staging System encompasses four stages. ARCO Stage I is the earliest stage of osteonecrosis and is characterized by a normal x-ray and an abnormal MRI. ARCO Stage IV is the most advanced stage of osteonecrosis and is characterized by findings of osteoarthritis on x-ray.
Change in Pain using the Pain VAS scale | Up to 24 months
  This is assessed using the pain Visual Analogue Scale (VAS). The participant marks an X on a 10cm scale denoting the level of pain that they are experiencing. VAS measures pain intensity on a scale of 0 (no pain) to 10 (worst pain).
Time to failure of femoral head | Up to 24 months
  Time is measured in months following the intervention (core decompression or core decompression with cells). Failure is defined as radiological progression to ARCO Stage III or IV or unremitting pain requiring surgical intervention.

SECONDARY OUTCOMES:
Change in Pain using the Hip disability and Osteoarthritis Outcome Score (HOOS) | Baseline, 6 months, 12 months, 24 months
  The Pain subscale of the Hip disability and Osteoarthritis Outcome Score (HOOS) will be used. The HOOS Pain sub-score is comprised of 10 items with a potential total of 40 points. Higher score worse pain,
Change in Symptoms and Stiffness using the HOOS | Baseline, 6 months, 12 months, 24 months
  The Symptoms and Stiffness will be assessed using the HOOS Symptoms and Stiffness sub-score is comprised of 5 items with a potential total score of 20 points. Higher score worse stiffness.
Change in Activities of Daily Living function using the HOOS | Baseline, 6 months, 12 months, 24 months
  The HOOS Activities of Daily Living function sub-score is comprised of 17 items with a potential total of 68 points. Higher scores better functioning.
Change in Function in Sports and Recreational Activities using the HOOS | Baseline, 6 months, 12 months, 24 months
  The HOOS Function of Sports and Recreational Activities subscale is comprised of 4 items with a potential total of 16 points. Higher score better outcome.
Change in Quality of Life using the HOOS | Baseline, 6 months, 12 months, 24 months
  The HOOS Quality of Life subscale is comprised of 4 items with a potential total of 16 points. Higher score better quality of life.
Change in Mental Health Composite Score using the PROMIS 10 Global Health Questionnaire | Baseline, 6 months, 12 months, 24 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) 10 Global Questionnaire is a 10-item patient-reported outcomes measure. A Mental Health Composite Score is generated as a summary of 4 items. Item responses range from 5 = None to 1 = Very Severe. The raw scores are converted into a T-score. Range 0 - 100; Population mean 50, standard deviation 10.
  PROMIS mental health survey. The measures are generic, rather than disease-specific, and use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. It is a survey of 10 questions which gives a physical health and mental health score. The raw global health mental score (4-20) is converted to a mental health T score (16.2-67.7). The higher the score, the better the health outcome.
Change in Physical Health Composite Score using the PROMIS 10 Global Health Questionnaire | Baseline, 6 months, 12 months, 24 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) 10 Global Questionnaire is a 10-item patient-reported outcomes measure. A Physical Health Composite Score is generated from the PROMIS 10 Global Questionnaire as a summary of 4 items. Item responses range from 5 = None to 1 = Very Severe. The raw scores are converted into a T-score. Range 0 - 100; Population mean 50, standard deviation 10.
  PROMIS physical health survey. The measures are generic, rather than disease-specific, and use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. It is a survey of 10 questions which gives a physical health and mental health score. The raw global health physical score (4-20) is converted to a physical health T score (16.2-67.7). The higher the score, the better the health outcome.
Change in Activity using the University of California Los Angeles (UCLA) Activity Rating Scale | Baseline, 6 months, 12 months, 24 months
  The UCLA Activity Score ranks the level of participant activity on a 10-point scale based on descriptors of activity ranging from wholly inactive and dependent on others, cannot leave residence (Level 1) to regular participation in impact sports such as tennis, skiing, acrobatics, ballet, heavy labor, or backpacking (Level 10). The higher the level, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne C Jones, PhD, Principal Investigator — Johns Hopkins University; Michael A Mont, MD, Principal Investigator — Sinai Hospital of Baltimore / LifeBridge Health; Stuart B Goodman, MD, PhD, Principal Investigator — Stanford University
Locations (10):
- United States (10):
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health Orthopedic Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be performed in accordance with the NIH Data Sharing Policy and Guidance document.
Supporting Information: CSR
Time Frame: In agreement with the policy of the National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), the data will be shared within 2 years after posting of the study results.
Access Criteria: 1. Clinicians and scientists will submit final peer-reviewed journal manuscripts. The public will have access to the published results.
  2. Requests for subsets of data for sub-analysis will be provided to all Co-Principal Investigators and Co- Investigators following approval of a submitted proposal.
  3. A limited access data (LAD) program for public access to a subset of de-identified data from our study will be developed, complying with all the data elements defined by the Health Insurance Portability and Accountability Act of 1996.
URL: https://sharing.nih.gov/data-management-and-sharing-policy